CLINICAL TRIAL: NCT04705610
Title: EYE-SEP : Study of Social Cognition in Patients With Multiple Sclerosis, From a Study of Eye Movement and Gaze Strategies Using Video-oculography.
Brief Title: Social Cognition in Multiple Sclerosis, From a Study of Eye Movement and Gaze Strategies Using Video-oculography
Acronym: EYE-SEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association de Recherche Bibliographique pour les Neurosciences (Other)
Collaborators: Centre Hospitalier Universitaire de Nice (Other); Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EYE-SEP
Record Dates: First submitted 2021-01-06; First posted 2021-01-12 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Multiple Sclerosis (MS); Multiple Sclerosis (MS) Relapsing Remitting; Multiple Sclerosis (MS) Primary Progressive; Multiple Sclerosis (MS) Secondary Progressive; Radiologically Isolated Syndrome; Clinically Isolated Syndrome; Healthy
Keywords: Demyelinating disease; Video-oculography; Eye-Tracking; Visual exploration strategies; Oculomotor behaviors; Oculomotor disorders; Emotions recognition; Social behavioral disorders; Social cognition; brain MRI
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Demyelinating Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, descriptive, comparative (case-control), monocentric study. Control are healthy volunteers. Pathological groups are Radiologically Isolated Syndrome (RIS), Clinically Isolated Syndrome (CIS), Relapsing-Remitting MS (RRMS), Secondary Progressive MS (SPMS) and Primary Progressive MS (PPMS).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Radiologically Isolated Syndrome (RIS) (Experimental)
  Interventions: Other: Video-oculography / Social cognition tasks / Neuropsychological evaluations
- Clinically Isolated Syndrome (CIS) (Experimental)
  Interventions: Other: Video-oculography / Social cognition tasks / Neuropsychological evaluations
- Relapsing-Remitting MS (RRMS) (Experimental)
  Interventions: Other: Video-oculography / Social cognition tasks / Neuropsychological evaluations
- Secondary Progressive MS (SPMS) (Experimental)
  Interventions: Other: Video-oculography / Social cognition tasks / Neuropsychological evaluations
- Primary Progressive MS (PPMS) (Experimental)
  Interventions: Other: Video-oculography / Social cognition tasks / Neuropsychological evaluations
- Healthy volunteer (Experimental)
  Interventions: Other: Video-oculography / Social cognition tasks / Neuropsychological evaluations

INTERVENTIONS:
Other: Video-oculography / Social cognition tasks / Neuropsychological evaluations — * Recording of eye movements with a video-oculography device during oculomotor paradigms (Fixations, horizontal and vertical reflex saccades, horizontal and vertical smooth pursuit, anti-saccades)
  * Recording of eye gaze with a video-oculography device during emotions recognition tasks (Reading the Mind in the Eyes test (Baron-Cohen 2001); Ekman Faces task (1976))
  * Neurological evaluation
  * Neuropsychological evaluations
  * Social cognitions tasks
  * Behaviour assessment

SUMMARY:
This study aims to:

* analyze prospectively the prevalence of subclinical oculomotor disorders (OMDs) in different phenotypes of Multiple Sclerosis (MS) and to study correlations with brain MRI T2 data.
* highlight link between modification of visual exploration strategies to decode emotions, and social behavioral disorders, in patients with demyelinating disease, from early to clinically definite stages.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female.
* 18 years old and above.
* Sufficient written and oral expression in French.
* Covered by a health insurance system
* Written informed consent signed by the patient.
* For the MS group:

  * Patient diagnosed according to diagnostic criteria established by Polman et al. (2010): Radiologically Isolated Syndrome compatible with MS (RIS), Clinically Isolated Syndrome compatible with MS (CIS), Relapsing-Remitting MS, Secondary Progressive MS, or Primary Progressive MS.

  * Hospitalized or coming to perform a consultation.
* For the control group: No cognitive impairment (non pathological Mini-Mental State Examination (MMSE), according to age, gender and socio-cultural level).

Exclusion Criteria:

* General anaesthesia within 3 months.
* Ophthalmological problems preventing a video-oculography examination.
* Oculomotor disorders:

  * For the control group: "fixation disorders" or "ocular tracking disorders".
  * For the MS group: atypical disorders.
* Cognitive disorders of the type: visual agnosia, visuo-spatial disorder, visuo-perceptual disorder or aphasia.
* Other neurological or ophthalmological disorders than MS
* History of stroke.
* Psychotropic drugs consummation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Prevalence of Oculomotor disorders (OMD) | Day 0
  To analyze prevalence of OMD in different MS phenotypes Eye movements were recorded and analyzed with an eye-tracking device during oculomotor paradigms (Fixations, horizontal and vertical reflex saccades, smooth pursuit and anti-saccades). For each subject values were judged abnormal if they differed by >1.65 Standard Deviation (SD) compared to their reference sample.
Eye gaze strategies during Emotion recognition: Affective Theory of Mind (ToM) | Day 0
  Comparison of gaze patterns between control group and pathological groups, during Affective ToM task. Evaluation criteria: number and duration of fixations. Eye movements were recorded with an eye-tracking device. Affective ToM was assessed using the " Reading the Mind in the Eyes " test (Baron-Cohen 2001).
Eye gaze strategies during Emotion recognition assessment: Facial emotion recognition (FER) | Day 0
  Comparison of gaze patterns between control group and pathological groups, during Facial emotion recognition tasks. Evaluation criteria: number and duration of fixations on areas of interest. Eye movements were recorded with an eye-tracking device. FER was assessed using some pictures from the Ekman Faces task (1976).

SECONDARY OUTCOMES:
T2 MRI lesion location: Posterior fossa lesions | Day 0
  T2 MRI performed by subjects in routine care. MRI data were described according to their nature (Posterior fossa lesions/ Brainstem-Cerebellum), and classified as present or absent. This is used for correlation study with Oculomotor disorders.
T2 MRI lesion location: Spinal cord lesions | Day 0
  T2 MRI performed by subjects in routine care. MRI data were described according to their nature, and classified as present or absent. This is used for correlation study with Oculomotor disorders.
T2 MRI lesion location: T2 lesions load | Day 0
  T2 MRI performed by subjects in routine care. MRI data were described according to their nature (>9T2), and classified as present or absent. This is used for correlation study with Oculomotor disorders.
Oculomotor paradigms raw performance - Horizontal saccades | Day 0
  This concerns saccades Latency (in ms), Main velocity (in °/sec) and Gain (gaze accuracy) during horizontal paradigms. Eye movements were recorded and analyzed with an eye-tracking device. These outcome measures are used in correlation and comparison analysis.
Oculomotor paradigms raw performance - Vertical saccades | Day 0
  This concerns saccades Latency (in ms), Main velocity (in °/sec) and Gain (gaze accuracy) during vertical paradigms. Eye movements were recorded and analyzed with an eye-tracking device. These outcome measures are used in correlation and comparison analysis.
Disease Disability | Day 0
  Disease Disability is assessed with the Expanded Disability Status Scale (EDSS), method of quantifying disability in multiple sclerosis. The EDSS scale ranges from 0 to 10 in 0,5-unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist. EDSS is used among other things for correlation study with Oculomotor disorders and oculomotor paradigms raw performance.
Disease Duration | Day 0
  Disease duration corresponds to years of evolution since initial diagnosis of the disease. It is based on an interview with subject's neurologist, or subject's medical file. Disease duration is used among other things for correlation study with Oculomotor disorders and oculomotor paradigms raw performance.
Correlations between visual exploration strategies and behavioral disorders. | Day 0
  To study correlations between gaze patterns and Neuropsychiatric Inventory (NPI). Evaluation criteria: number and duration of fixations on areas of interest during social cognition task (" Reading the Mind in the Eyes " test (Baron-Cohen 2001) and Ekman Faces task). Eye movements were recorded with an eye-tracking device. Behavior disorders were assessed with the Neuropsychiatric Inventory.
Correlations between visual exploration strategies and social cognition impairment: Facial emotion recognition. | Day 0
  To study correlations between gaze patterns and Facial emotion recognition tasks. Evaluation criteria: number and duration of fixations on areas of interest during Facial emotion recognition tasks (Ekman Faces task). Eye movements were recorded with an eye-tracking device. Facial emotion recognition impairment with the Ekman Faces task.
Correlations between visual exploration strategies and social cognition impairment: Affective ToM. | Day 0
  To study correlations between gaze patterns and Affective ToM. Evaluation criteria: number and duration of fixations during " Reading the Mind in the Eyes " test (Baron-Cohen 2001)). Eye movements were recorded with an eye-tracking device. Affective ToM impairments with the " Reading the Mind in the Eyes " test (Baron-Cohen 2001).
Correlations between Facial emotion recognition and behavioral disorders. | Day 0
  To study correlations between Facial emotion recognition tasks and Neuropsychiatric Inventory (NPI). Evaluation criteria: Ekman scores and NPI scores. Behavior disorders were assessed with the Neuropsychiatric Inventory.
Correlations between Emotion recognition and behavioral disorders. | Day 0
  To study correlations between Affective ToM task and Neuropsychiatric Inventory (NPI). Evaluation criteria: " Reading the Mind in the Eyes " scores (Baron-Cohen 2001). Behavior disorders were assessed with the Neuropsychiatric Inventory.
Correlations between Facial emotion recognition and disability level. | Day 0
  To study correlations between Facial emotion recognition tasks and Expanded Disability Status Scale (EDSS). Evaluation criteria: Ekman scores and EDSS scores.
Correlations between Emotion recognition and disability level. | Day 0
  To study correlations between Affective ToM task and Expanded Disability Status Scale (EDSS). Evaluation criteria: " Reading the Mind in the Eyes " scores (Baron-Cohen 2001).
  Disability level were assessed with the Expanded Disability Status Scale.
Correlations between Cognitive Theory of mind and disability level. | Day 0
  To study correlations between Cognitive Theory of mind task and Expanded Disability Status Scale (EDSS). Evaluation criteria: TOM-15 scores (TOM-15 a false-belief task to assess cognitive theory of mind). Disability level were assessed with the Expanded Disability Status Scale.
Correlations between Affective empathy and disability level. | Day 0
  To study correlations between Affective empathy and Expanded Disability Status Scale (EDSS). Evaluation criteria: The Empathy Quotient (EQ) scores. Disability level were assessed with the Expanded Disability Status Scale.
Eye gaze strategies during exploration of a specific artwork | Day 0
  Comparison of gaze patterns between control group and pathological groups, during exploration of a specific artwork. Evaluation criteria: difference in exploration strategy (chronology) on target areas.

CONTACTS AND LOCATIONS:
Overall Officials: Christine LEBRUN-FRENAY, PUPH, Principal Investigator — Centre de Ressources et de Compétences SEP, UMRC Pasteur 2, Université Nice Côte d'Azur, Nice-France; Alain PESCE, PUPH, Principal Investigator — Centre Mémoire, Centre de Gérontologie Clinique RAINIER III, Princess Grace Hospital (Monaco); Benoit KULLMANN, MD-PHD, Study Director — AREBISN (Association de Recherche Bibliographique pour les Neurosciences), Nice (France)
Locations (1):
- Centre Mémoire / Centre de Gérontologie Clinique Rainier III / Princess Grace Hospital, Monaco, Monaco

REFERENCES:
- See also: K. Polet, et al.. Video-oculography in multiple sclerosis: Links between oculomotor disorders and brain magnetic resonance imaging (MRI). Multiple Sclerosis and Related Disorders, 2020-05-01, Volume 40, Article 101969 — https://doi.org/10.1016/j.msard.2020.101969